CLINICAL TRIAL: NCT06528912
Title: Standard Follow-up Program (SFP) for Neuro-oncology Cancer Patients Treated With Radiotherapy
Brief Title: Standard Follow-up Program Neuro-oncology Patients (SFP Neuro-Oncology)
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: SFP Neuro-Oncology
Record Dates: First submitted 2024-02-26; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Neurological Cancer
Keywords: Acute toxicity; Late toxicity; Prediction models
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Radiotherapy — Follow-up

SUMMARY:
Standardised evaluation of baseline data regarding tumor-, patient- and treatment-characteristics as well as follow-up data regarding tumor- and clinical-outcome of neuro-oncology patients treated with radical/curative radiotherapy.

Motive:

Currently there is limited data on dose-effect relationships of tissues and structures in and around the brain. This lack of knowledge hampers patient selection for proton therapy, technique innovations, and accurate prediction of treatment outcome.

Goal:

To evaluate the selection for radiation treatment, obtain more knowledge on dose-effect relationships and enable insight in necessary treatment technique innovations that would improve treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patient with neuro-oncological cancer
* Patient receiving a radiotherapy dose XXX Gy

Exclusion Criteria:

* Failure to comply with any of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: neuro-oncology patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2040-01 (Estimated); Study Completion 2040-01 (Estimated)

PRIMARY OUTCOMES:
Treatment associated CNS toxicity | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Treatment associated CNS Toxicity
Radionecrosis | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Treatment associated radionecrosos measured with CTCAE

SECONDARY OUTCOMES:
Treatment associated non-CNS toxicity | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy
  Treatment associated non-CNS toxicity
Overall survival | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Overall survival
Progression free survival | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy
  Progression free survival

OTHER OUTCOMES:
Patient-rated Quality of Life | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Patient-rated quality of Life is measured with the Quality-of-Life Questionnaire-C30 (EORTC QLQ-C30)
Patient-rated Quality of Life | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Patient-rated quality of Life is measured with the Quality-of-Life Questionnaire Brain Cancer module (EORTC QLQ-BN20)
Patient-rated Quality of Life | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Patient-rated quality of Life is measured with the EuroQol Health questionnaire 5-level version (EuroQoL-5D-5L)
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Patient-rated cognition is measured with the Groninger Cognitionlist (GroCo)
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Rey's auditory verbal learning test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Doors test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Semantic fluency test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Boston naming test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Controlled oral word association test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Trail making test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Digit span test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Symbol digit modality test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Vienna test system test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the FEEST test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Key search test
Cognition | Before start of radiation therapy, at 2,5 years; 5 years 7,5 years, 10 years and 12,5 years after completion of radiation therapy.
  Cognition measured with the Zoo map test

CONTACTS AND LOCATIONS:
Locations (1):
- UMCG, Groningen, Netherlands